CLINICAL TRIAL: NCT07335341
Title: Case-Specific Health Care Professional Clinical Survey of Liberant™ Thrombectomy System
Status: Not yet recruiting | Type: Observational
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT25034
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Venous Embolism of Lower Extremities (Diagnosis); Arterial Embolism and Thrombosis; Acute DVT of Lower Extremity; Chronic DVT of Lower Extremity; DVT; Deep Vein Thrombosis Leg; Thrombus in the Peripheral Venous Vasculature; Peripheral Arterial Disease; Acute Limb Ischemia; Lower Extremity Acute Limb Ischemia; LE ALI
Keywords: Thrombus in Peripheral Arterial Systems; Thrombectomy; Thrombosis; Venous Thrombosis; Aspiration Thrombectomy; Percutaneous Mechanical Thrombectomy; Arterial Occlusive Diseases; Vascular Diseases; Peripheral Vascular Diseases; Peripheral Arterial Disease; Mechanical Thrombectomy; Aspiration; Liberant Thrombectomy System; adverse events; Excipio; Thrombus in Peripheral Venous Systems
MeSH Terms: conditions — Disease; Thrombosis; Venous Thrombosis; Peripheral Arterial Disease; Arterial Occlusive Diseases; Vascular Diseases; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Liberant Thrombectomy System — The Liberant thrombectomy system is indicated for the removal of fresh, soft emboli or thrombi from the vessels of the peripheral arterial and venous systems

SUMMARY:
The purpose of Case-Specific Health Care Professional (HCP) Clinical Survey of Liberant™ Thrombectomy System, also known as the Liberant Clinical Assessment, is to collect first-in-human clinical data to confirm the safety and performance of the Medtronic Liberant™ thrombectomy system when used for the removal of fresh, soft emboli or thrombi from the vessels of the peripheral arterial and venous systems

DETAILED DESCRIPTION:
The Liberant Clinical Assessment is a multicenter, prospective per patient HCP recollection survey. Participating HCPs will document their individual case experience following routine utilization of Liberant in accordance with the approved device labeling. Individual use cases will be entered within 72 hours of device usage to identify periprocedural incidents of risk and evaluate device performance. At least 50 use cases will be collected and aggregated from at least 10 participating HCPs. This data collection is for a single point in time, with no patient follow-up. Individual HCP responses for each case will be aggregated by a third party vendor.

ELIGIBILITY:
Patient case selection to be included in the clinical assessment will be specific to Liberant and will be made according to the following criteria:

1. Patient treated is age ≥ 22 years at the time of procedure
2. Use of Liberant in accordance with the device labeling within 72 hours of index procedure

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Liberant thrombectomy system is intended for use in adult patients with occluded peripheral arterial and venous vessels.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of Device related Serious Adverse Event at Index procedure | Index Procedure
  An Adverse Event that converted to Serious Adverse Event, involving the function of the subject device, or the presence of the device in the body, including events that are directly attributable to the Liberant Thrombectomy System
Rate of technical success at Index procedure | Index procedure
  Technical success: Successful introduction, delivery, aspiration of fresh, soft emboli or thrombi, and retrieval of the Liberant per the Instructions for Use (IFU) during the index procedure
Rate of Procedural Success at Index procedure | Index procedure
  Procedure success: Successful removal of fresh, soft emboli or thrombi and restoration of adequate blood flow, inclusive of all endovascular therapies during the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: John R Laird Jr, MD, Principal Investigator — Medtronic Endovascular

IPD SHARING:
Plan to Share IPD: No
No patients will be engaged, and no medical records will be accessed or used. Individual HCP responses for each case will be aggregated into a final report.